CLINICAL TRIAL: NCT00132990
Title: A Multicenter Pilot Study of Pallidal Deep Brain Stimulation of Cervical Dystonia
Brief Title: A Multicenter Pilot Study of Pallidal Deep Brain Stimulation for Cervical Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Calgary Health Region (Other); Medtronic (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16760
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2007-01

CONDITIONS: Cervical Dystonia
Keywords: Cervical dystonia; Deep brain stimulation
MeSH Terms: conditions — Torticollis | interventions — Deep Brain Stimulation

INTERVENTIONS:
Device: Deep brain stimulation

SUMMARY:
The purposes of this study are:

* to determine if bilateral pallidal deep brain stimulation results in improvement in neck postures/movements;
* to determine if bilateral pallidal deep brain stimulation results in improvement in quality of life; and
* to document the adverse effects of surgery in patients with cervical dystonia.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the globus pallidus has been proposed as a treatment for cervical dystonia. At present there are only anecdotal reports of benefit. The objective of this project is to prospectively assess the outcomes of DBS on cervical dystonia in a blinded manner. Our hypothesis is that in patients refractory to medical management, bilateral pallidal DBS will reduce the severity of cervical dystonia at 1 year follow up.

The research plan is that of a feasibility study, examining outcomes of 10 patients who would be referred for surgical management due to the severity of their disease. The Toronto Western Spasmodic Torticollis Rating Scale (TWSTR) will be preformed by a blinded neurologist at the completion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female
* Diagnosed with cervical dystonia by a movement disorders neurologist
* Has cervical dystonia alone, not generalized or multifocal
* Has had adequate trials of medical therapy

Exclusion Criteria:

* Cognitive impairment
* Abnormalities on pre-operative magnetic resonance imaging (MRI)
* Medical conditions precluding general anaesthetic or surgery
* Unstable psychiatric disease
* Previous brain lesions to treat cervical dystonia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-02; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Improvement in neck postures/movements
Improvement in quality of life

SECONDARY OUTCOMES:
Document adverse effects of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zelma Kiss, MD, Principal Investigator — University of Calgary
Locations (5):
- Canada (5):
  - Dr. Zelma Kiss, Calgary, Alberta
  - Dr. Matt Wheatley, Edmonton, Alberta
  - Dr. Chris Honey, Vancouver, British Columbia
  - Dr. Jerry Krcek, Winnipeg, Manitoba
  - Dr. Andrew Parrent, London, Ontario

REFERENCES:
- [Derived] Kiss ZH, Doig-Beyaert K, Eliasziw M, Tsui J, Haffenden A, Suchowersky O; Functional and Stereotactic Section of the Canadian Neurosurgical Society; Canadian Movement Disorders Group. The Canadian multicentre study of deep brain stimulation for cervical dystonia. Brain. 2007 Nov;130(Pt 11):2879-86. doi: 10.1093/brain/awm229. Epub 2007 Sep 28. PMID 17905796
- See also: Related Info — http://www.wemove.org
- See also: Related Info — http://www.medtronic.com